CLINICAL TRIAL: NCT01067378
Title: Peer Debriefing Versus Instructor Debriefing for Interprofessional Simulation Based Education (PICS
Brief Title: Peer Debriefing Versus Instructor Debriefing for Interprofessional Simulation Based Education
Acronym: PICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SMH09172
Record Dates: First submitted 2010-02-01; First posted 2010-02-11 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Crisis Resource Management
Keywords: Interdisciplinary Health Team; Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expert instructor debriefing (Active Comparator): Expert instructor debriefing
  Interventions: Other: Expert instructor debriefing
- Peer-led debriefing (Experimental): Peer-led debriefing
  Interventions: Other: Peer-led debriefing

INTERVENTIONS:
Other: Peer-led debriefing
  Arms: Peer-led debriefing
Other: Expert instructor debriefing
  Arms: Expert instructor debriefing

SUMMARY:
Crisis management is important for operating room practice and non-technical skills are acknowledged as key to ensure patient safety in these situations. Unfortunately, it can be difficult to find instructors with appropriate experience. A peer-led team debriefing is led by the team it self rather than an external expert instructor but remains a reflective process. Incorporating peer-led debriefing compared to expert-led debriefing may increase access to an interprofessional crisis resource management course using simulation.

The goals of the study are to observe the effect of an interprofessional peer-led team debriefing in the change in performance of non-technical skills of team performance and to compare it with the "gold standard" of expert-led debriefing on the performance of non-technical skills during a simulated operating room crisis.

The investigators hypothesize that interprofessional peer-led debriefing will improve the performance of non-technical skills of the team during simulated intraoperative crisis management and that this improvement will be equivalent to the "gold standard" expert-led debriefing.

ELIGIBILITY:
Inclusion Criteria:

* Operating room (OR) nurses from St. Michael's Hospital and University of Toronto Anesthesia and Surgery Residents/Fellows

Exclusion Criteria:

* OR nurses from other hospitals and Residents/Fellows from other programs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Performance of non-technical skills of the teams. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Allan Waters' Family Patient Simulation Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Boet S, Bould MD, Sharma B, Revees S, Naik VN, Triby E, Grantcharov T. Within-team debriefing versus instructor-led debriefing for simulation-based education: a randomized controlled trial. Ann Surg. 2013 Jul;258(1):53-8. doi: 10.1097/SLA.0b013e31829659e4. PMID 23728281